CLINICAL TRIAL: NCT01498549
Title: Cognitive Effects of Atomoxetine in Humans: Genetic Moderators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Prinicipal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1103008235
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Addiction
Keywords: Abstinent cocaine users; cognitive testing
MeSH Terms: conditions — Behavior, Addictive | interventions — Atomoxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Active Comparator): Atomoxetine compared to the sugar pill
  Interventions: Drug: Sugar Pill
- Sugar Pill (Placebo Comparator): Sugar pill compared to atomoxetine
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine 40mg and 80mg compared to the sugar pill
  Other Names: Strattera
  Arms: Sugar Pill
Drug: Sugar Pill — Sugar pill compared to Atomoxetine 40mg and 80mg.
  Other Names: placebo
  Arms: Atomoxetine

SUMMARY:
The overall goal of this study is to determine if atomoxetine treatment improves selective cognitive functions in abstinent cocaine users, compared to healthy controls. The study will also test if a functional variation of the NET promoter polymorphic region (NETpPR) moderates the cognitive effects of atomoxetine.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled, crossover study, with cocaine use (cocaine users vs. healthy controls) and NET AAGG4 status (L4/ L4 vs. L4/S4 or S4/ S4 genotype) as the between-subject factors. Similar to previous studies, we propose to compare individuals with two copies of the L4 allele to participants with at least one S4 allele because only less than two percent of the general population is homozygous for the S4 allele. Forty cocaine users and 40 healthy controls will participate in 3 test sessions, where they will be assigned to 40 mg atomoxetine, 80 mg atomoxetine, or placebo. Outcome measures will include physiological, subjective, and cognitive performance measures.

To date this study has 35 completers and currently in data analysis. (January 2016)

ELIGIBILITY:
Inclusion Criteria:

* Male and females, between the ages of 21 and 50;
* No current dependence or abuse of drugs of abuse or alcohol (except and tobacco);
* No current medical problems and normal ECG;
* For women, not pregnant as determined by pregnancy screening nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* Current major psychiatric illnesses including mood, psychotic, or anxiety disorders;
* History of major medical illnesses; including liver diseases, heart disease, or other medical conditions that the physician investigator deems contraindicated for the subject to be in the study;
* Known allergy to Atomoxetine;
* Use of Monoamine Oxidase inhibitor within the last month (clinically Atomoxetine administration is contraindicated with or within 2 weeks of discontinuation of Monoamine oxidase inhibitor therapy).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Participants were randomly assigned to one of 3 possible groups over a 3 day assessment period.
Period: Overall Study
Arm/Group | Participants
Started | 39
Atomoxetine 40 mg | 39
Atomoxetine 80 mg | 37
Sugar Pill 0 mg | 36
Completed (Completed all 3 days for each arm in the crossover design.) | 35
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: The total number of people enrolled in the study before randomization to crossover assignment.
Groups:
- Total Sample: This is the summary of the total sample used in the crossover design.
Arm/Group | Total Sample
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.21 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rapid Visual Information Processing
Description: Cognitive Test to determine the speed of Visual information. The CANTAB Rapid Visual Information Processing test (RVP) is a measure of sustained attention with a small working memory component (Sahakian and Owen, 1992). Digits are rapidly (100/minute) and pseudo-randomly presented for 7 minutes. Subjects are instructed to press when the third digit of a target sequence (e.g. 3-5-7) is displayed. Primary outcomes are indices of target discriminability (A') and response bias (B") and response latency to targets.
Time Frame: 2 years
Population: Participants that completed any arm in the crossover are included in the analysis.
Measure: Mean (Standard Deviation); unit: Proportion of Participants
Groups:
- Atomoxetine 40 mg: Atomoxetine 40 mg dose
- Atomoxetine 80 mg: Atomoxetine 80 mg dose
- Sugar Pill 0mg: Sugar pill 0mg dose
Arm/Group | Atomoxetine 40 mg | Atomoxetine 80 mg | Sugar Pill 0mg
Number analyzed (Participants) | 39 | 37 | 36
Proportion of Participants
  Descriminability | 0.88 (0.06) | 0.89 (0.07) | 0.87 (0.05)
  Response Bias | 0.87 (0.14) | 0.86 (0.16) | 0.89 (0.22)

2. Primary Outcome: Rapid Visual Information Processing: Mean Correct Response Latency
Description: as for outcome 1
Time Frame: 2 years
Population: Participants that completed any arm in the crossover are included in the analysis, participants with valid observations at both indices are included in the calculation.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Sugar Pill 0mg: Sugar pill 0 mg dose
Arm/Group | Atomoxetine 40 mg | Atomoxetine 80 mg | Sugar Pill 0mg
Number analyzed (Participants) | 38 | 37 | 36
milliseconds | 446.70 (106.84) | 452.64 (133.22) | 464.44 (113.07)

ADVERSE EVENTS:
Time Frame: Adverse events were collected once for each of the three visits on all enrolled subjects.
Description: The assessment of adverse events utilized the Brief Symptom Inventory (BSI), an instrument that consists of 77 items.
Groups:
- Sugar Pill 0 mg: Sugar pill 0 mg dose
Arm/Group | Atomoxetine 40 mg | Atomoxetine 80 mg | Sugar Pill 0 mg
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 1/39 | 1/39 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine 40 mg (N=39) | Atomoxetine 80 mg (N=39) | Sugar Pill 0 mg (N=39)
nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
other (General disorders) | 1 (1) | 0 (0) | 1 (1) — non-life threatening, non-specific event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes